CLINICAL TRIAL: NCT05843097
Title: SnapSBO - An International Non-randomized Time-bound Prospective Observational Cohort Study Addressing the Epidemiology and Management of Small Bowel Obstruction
Brief Title: SnapSBO - Small Bowel Obstruction Snapshot Audit
Acronym: SnapSBO
Status: Completed | Type: Observational
Sponsor: European Society for Trauma and Emergency Surgery (Other)
Responsible Party: Principal Investigator, Isidro Martinez Casas, MD PhD, Chair, SnapSBO Steering Group, European Society for Trauma and Emergency Surgery
Other Study IDs: ESTESSnapSBO202324
Record Dates: First submitted 2023-03-10; First posted 2023-05-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Small Bowel Obstruction
Keywords: diagnosis; management; guidelines; outcomes
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Small bowel obstruction (SBO) and its complications are frequently seen in patients admitted through the Emergency Departments of all acute care hospitals2.

There is variation in the optimal use of imaging, the appropriate timing and duration of non-operative management attempts, anti-microbial therapies, and the criteria for surgical management, which results in heterogeneity in approaches and outcomes across international clinical centers. The expected number of SBO cases in most clinical centers is predictable, enabling a suitably-sized cohort of patients to be gathered in the snapshot audit.

This 'ESTES snapshot audit' -a prospective observational cohort study- has a dual purpose. Firstly, as an epidemiological study, it aims to uncover the burden of disease. Secondly, it aims to demonstrate current strategies employed to diagnose and treat these patients. These twin aims will serve to provide a 'snapshot' of current practice, but will also be hypothesis-generating while providing a rich source of patient-level data to allow further analysis of the particular clinical questions.

DETAILED DESCRIPTION:
Prospective audit of consecutive patients admitted in Emergency Department for mechanical small bowel obstruction over a 3-month period. The audit shall include unscheduled patient admissions from November 2023 until May 2024 as outlined in 'Key Study Dates'.

As this is an observational cohort audit, no change to normal patient management is required.

Primary Objective

To explore differences in patients, management and outcomes across the entire cohort to identify areas of practice variability resulting in apparent differences in outcome warranting further study. The outcomes that the study will examine are:

* Incidence of small bowel obstruction by etiology.
* Differences in clinical presentation.
* Diagnostic work-up.
* Non-operative management strategies.
* Time to surgery and outcomes.
* Complications related to disease and/or therapies within 60 post-operative days.
* Length of Emergency Department and Hospital stay.
* Re-admission within 6 months for related conditions.

Methods for identifying patients

Multiple methods may be used according to local circumstances/staffing:

1. Daily review of emergency department (non-operative) and operating room lists.
2. Daily review of team handover sheets / emergency admission lists / ward lists.
3. Review of operating room logbooks.
4. Use of electronic systems to flag any readmissions of patients identified and treated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥16 years of age) admitted for mechanical small bowel obstruction. Example etiologies which should be included:

  1. Adhesions.
  2. Hernias with bowel compromise (incisional/parastomal, ventral, inguinal, femoral, obturator, internal).
  3. Malignancy (primary: lymphoma, carcinoid, GIST, adenocarcinoma/metastatic disease: colon, ovarian, gastric, pancreatic, melanoma and others).
  4. Enteroliths/gallstones/bezoars/foreign bodies
  5. Radiation.
  6. Inflammation (Crohn's disease, mesenteric adenitis, appendicitis, diverticulitis, tuberculosis, actinomycosis, ascariasis).
  7. Congenital (malrotation, duplication cysts).
  8. Trauma (hematomas, ischemic strictures).

Exclusion Criteria:

* Functional small bowel obstruction (dysmotility or adynamic ileus secondary to abdominal operations, peritonitis, trauma or medications).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients (≥16 years of age) admitted for mechanical small bowel obstruction.
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Small Bowel Obstruction, by etiology | 6 months
  This study aims to quantify (as an integer, n) the etiologies of small bowel obstruction (adhesions, hernias, malignancy and other causes)
Time to Surgical Treatment of Small Bowel Obstruction vs Outcomes | 6 months
  Time (hours) from hospital admission to Surgical Treatment of Small Bowel Obstruction vs Outcomes

SECONDARY OUTCOMES:
Complications related to operative or non-operative management of small bowel obstruction | 6 months from hospital admission
  Complications related to operative or non-operative management of small bowel obstruction (integer count n,%) - for example haemorrhage, wound infection, venous thromboembolism, anastomotic leak
Adherence to evidence-based guidelines vs outcomes | 6 months from hospital admission
  Adherence to evidence-based World Society of Emergency Surgery Bologna guideline 2020 recommendations (Table 5: available here https://wjes.biomedcentral.com/articles/10.1186/s13017-018-0185-2/tables/5) vs outcomes (30-day post operative or hospital discharge survival (median days), length of hospital stay (median days), Complications related to operative or non-operative management of small bowel obstruction (integer count n,%) - for example haemorrhage, wound infection, venous thromboembolism, anastomotic leak (integer count n,%)
Patient-related Outcome Metrics for Surgical vs Non-operative management | At first post-discharge clinic visit, anticipated within 6 months of admission
  Patient-related Outcome Metrics for Surgical vs Non-operative management, using the PROdiGI (Patient Reported Outcome Measure for GastroIntestinal Recovery) qualitative quality-of-life assessment tool specifically designed for gastro-intestinal symptoms in adult patients undergoing major abdominal surgery for indications OR patients being treated for intestinal obstruction regardless of etiology. Patients will be assisted in completing an anonymous survey where domains of gastrointestinal function are assessed using a 20-element Likert scales (with higher scores denoting worse perceived function) and a Visual Analog Scale 0-100 grading function from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Isidro Martínez Casas, MD PhD, Principal Investigator — Hospital Universitario Virgen del Rocio
Locations (1):
- Hospital Universitario Virgen del Rocio, Seville, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The ESTES SnapAppy Group welcomes the use of these de-identified pooled data for further research that benefits patients. Requests can be submitted to the ESTES Research Committee. Release is subject to their approval and the appropriate safeguarding as determined by applicable legislation (GDPR and HIPAA).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After study main conclusions are published
Access Criteria: Being one of study participating centers investigators

REFERENCES:
- [Background] Bass GA, Kaplan LJ, Ryan EJ, Cao Y, Lane-Fall M, Duffy CC, Vail EA, Mohseni S. The snapshot audit methodology: design, implementation and analysis of prospective observational cohort studies in surgery. Eur J Trauma Emerg Surg. 2023 Feb;49(1):5-15. doi: 10.1007/s00068-022-02045-3. Epub 2022 Jul 15. PMID 35840703

DOCUMENTS (1):
  • Study Protocol (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT05843097/Prot_000.pdf